CLINICAL TRIAL: NCT02999126
Title: Slow Stepwise Propofol TCI Induction for Titration Anesthesia Maintenance
Acronym: (TITINDUC)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Hernan Boveri, MD, Hospital Italiano de Buenos Aires
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2884
Record Dates: First submitted 2016-12-08; First posted 2016-12-21 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Target Controlled Infusion; Induction of Anesthesia; Bispectral Index
Keywords: Total Intravenous Anesthesia; Titration; Target Controlled Infusion; Propofol; Bispectral index
MeSH Terms: interventions — Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Patients < 65 years old Propofol 1% TCI induction using plasma concentration, Marsh model (Ke0=0.26 min-1) at 1 mcg/ml, increasing the target concentration by 0.5 mcg/ml every minute until LOC. Remifentanil TCI 6 ng/ml and a neuromuscular relaxant will be administered afterwards in order to perform endotracheal intubation. CeLOC propofol concentration will be established and it will be observed for another 30 minutes. If BIS <40 or >65 propofol target concentration will be modified by 0,3 mcg/ml.
  Interventions: Drug: Propofol; Drug: Remifentanil Hydrochloride
- Group 2 (Experimental): Patients ≥ 65 years old Propofol 1% TCI induction using plasma concentration, Marsh model (Ke0=0.26 min-1) at 1 mcg/ml, increasing the target concentration by 0.5 mcg/ml every minute until LOC. Remifentanil TCI 6 ng/ml and a neuromuscular relaxant will be administered afterwards in order to perform endotracheal intubation. CeLOC propofol concentration will be established and it will be observed for another 30 minutes. If BIS <40 or >65 propofol target concentration will be modified by 0,3 mcg/ml.
  Interventions: Drug: Propofol; Drug: Remifentanil Hydrochloride

INTERVENTIONS:
Drug: Propofol — Propofol intravenously by a stepwise TCI titration with Marsh pharmacokinetic model
  Other Names: Fresofol
Drug: Remifentanil Hydrochloride — Remifentanil intravenously 6 ng/ml by TCI effect site, 3 min prior to intubation and maintained at that concentration throughout the study. If clinical signs of inadequate analgesia are present, remifentanil target concentration will be increased by 1 ng/ml.

SUMMARY:
The purpose of this study is to determine if a slow stepwise propofol TCI induction with Marsh model (Ke0 0.26), allows for an accurate estimation of the effect site concentration required for maintenance of the general anesthesia, with propofol and remifentanil, in adult populations older and younger than 65 years of age.

DETAILED DESCRIPTION:
Introduction: Currently, propofol is the most widely used intravenous anesthetic drug that is able to provide a safe general anesthesia. Propofol can be administered by using different techniques including target controlled infusion (TCI). The ability to maintain the pharmacological conditions after achieving a predetermined clinical effect is one of the major advantages of this technique. Although the use of TCI devices has increased in common clinical practice, whether or not all patients are suitable for TCI remains unclear. Pharmacological models were created based on information from healthy volunteers which may not apply for specific clinical conditions resulting either in over- or sub-dosed when using certain drugs.

It is not only individual variability in the pharmacokinetic (PK) parameters of the anesthetic that is a clinical problem, but it is also the pharmacodynamic variability. A previous study showed up to 6 times the inter-individual difference among young volunteers in loss of consciousness (LOC) and return of consciousness (ROC). In addition, greater differences may be found in the elderly.

Inaccurate general models require the anesthetic team to manually tailor medication requirements for each individual based on the desired therapeutic effect.

The purpose of this study is to evaluate if a slow stepwise propofol TCI induction with Marsh model (Ke0 0.26), assessed by clinical and electroencephalographic parameters, allows for an accurate estimation of the effect concentration required for hypnosis titration and maintenance of the general anesthesia, in adult populations older and younger than 65 years of age.

General Objective

• To establish whether a guided slow stepwise guided propofol induction with TCI represents a good correlation between the calculated Effect-Site Concentration (Ce) for the loss of consciousness and the required Ce to maintain a bispectral index (BIS) value between 45 and 65 during anesthesia maintenance in both age populations

Specific Objectives

* To determine the BIS value achieved with every propofol infusion based on the calculated Ce for the time of loss of consciousness (TLOC)
* To compare the drug infused per time unit required for the loss of consciousness in both groups
* To compare the time and Ce required to achieve loss of consciousness in both groups
* To evaluate the impact of remifentanil during hypnosis by using the BIS index

Hypothesis

During a slow stepwise anesthetic induction with TCI using the Marsh Model 4.0, the calculated Ce for the TLOC is comparable to the Ce required for the maintenance of the hypnosis during the general anesthesia, overcoming the inter-individual variability.

Methods

Experimental study, prospective clinical trial, phase 4. Each subject will be assigned to the propofol induction modality as described in the "intervention" section.

Once consciousness has been lost and maintenance target concentration has been established, manual ventilation will be initiated. Remifentanil TCI 6 ng/ml and a neuromuscular relaxant will be administered afterwards in order to perform endotracheal intubation. An infusion of phenylephrine between 0,1 and 0,4 mcg/kg/min will be initiated in order to maintain blood pressure values within 20% of the baseline value.

Continuous monitoring of BIS will be maintained after remifentanil infusion and intubation. Three minutes after endotracheal intubation, surgery will be prepared following standard procedures. BIS, spectrogram, and hemodynamics will be registered every 15 seconds, continuously, and every 3 minutes during 10 minutes respectively.

Subsequently, propofol Ce at TLOC will be established (if any modifications were necessary after TLOC) and it will be observed for another 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2.
* Age over 20 years old.
* Scheduled to undergo elective surgery of minor or medium complexity under general anesthesia.
* Regarding cognitive function: subjects will be considered with enough cognitive function if they are able to read and understand the medical history form by properly answering medical questions during the preoperative anesthesia assessment and being also able to sign the informed consent form.

Exclusion Criteria:

* Pregnancy.
* Obesity (BMI >30).
* Patients taking benzodiazepines or other central nervous system action drugs.
* Subjects with psychiatric disorders with or without treatment.
* Allergies or any adverse reaction to propofol or any of its components (egg lecithin).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Time that BIS range remains within 45 and 65 after a stepwise TCI titration | A 30-minute period, starting 10 minutes after Remifentanil infusion (when propofol and remifentanil plasma-effect compartment equilibration has been reached)
  TCI Effect Site Concentration achieved at LOC, depth of anesthesia will be recorded with BIS bilateral sensor

SECONDARY OUTCOMES:
Time for loss of consciousness | Up to First 10 minutes, from start of propofol infusion at time 0 until loss of verbal response
  In seconds, using TCI induction with Marsh 4.0 pharmacokinetic model
Effect Site Concentration required for loss of consciousness | Up to first 10 minutes. It will be considered the propofol effect site concentration displayed at the moment loss of consciousness is achieved.
  In mcg/ml, using Marsh Pharmacokinetic Model, Ke0 0.26 min-1

CONTACTS AND LOCATIONS:
Overall Officials: Hernán Boveri, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Struys M, Versichelen L, Byttebier G, Mortier E, Moerman A, Rolly G. Clinical usefulness of the bispectral index for titrating propofol target effect-site concentration. Anaesthesia. 1998 Jan;53(1):4-12. doi: 10.1111/j.1365-2044.1998.00279.x. PMID 9505735
- [Background] Coppens M, Van Limmen JG, Schnider T, Wyler B, Bonte S, Dewaele F, Struys MM, Vereecke HE. Study of the time course of the clinical effect of propofol compared with the time course of the predicted effect-site concentration: Performance of three pharmacokinetic-dynamic models. Br J Anaesth. 2010 Apr;104(4):452-8. doi: 10.1093/bja/aeq028. Epub 2010 Feb 26. PMID 20190259
- [Background] Bienert A, Wiczling P, Grzeskowiak E, Cywinski JB, Kusza K. Potential pitfalls of propofol target controlled infusion delivery related to its pharmacokinetics and pharmacodynamics. Pharmacol Rep. 2012;64(4):782-95. doi: 10.1016/s1734-1140(12)70874-5. PMID 23087131
- [Background] Iwakiri H, Nishihara N, Nagata O, Matsukawa T, Ozaki M, Sessler DI. Individual effect-site concentrations of propofol are similar at loss of consciousness and at awakening. Anesth Analg. 2005 Jan;100(1):107-110. doi: 10.1213/01.ANE.0000139358.15909.EA. PMID 15616062
- [Background] Struys MM, Sahinovic M, Lichtenbelt BJ, Vereecke HE, Absalom AR. Optimizing intravenous drug administration by applying pharmacokinetic/pharmacodynamic concepts. Br J Anaesth. 2011 Jul;107(1):38-47. doi: 10.1093/bja/aer108. Epub 2011 May 30. PMID 21624964
- [Background] Sepulveda PO, Cortinez LI, Recart A, Munoz HR. Predictive ability of propofol effect-site concentrations during fast and slow infusion rates. Acta Anaesthesiol Scand. 2010 Apr;54(4):447-52. doi: 10.1111/j.1399-6576.2009.02183.x. Epub 2009 Dec 14. PMID 20003124